CLINICAL TRIAL: NCT05135468
Title: A Multicenter, Randomized, Double-Blind, and Placebo-Controlled Phase 3 Clinical Study to Evaluate the Efficacy and Safety of Finasteride Spray (CU-40102) in Chinese Adult Male Patients With Androgenetic Alopecia (AGA)
Brief Title: A Phase 3 Clinical Study Patients With Androgenetic Alopecia (AGA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cutia Therapeutics（Wuxi）Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CU-40102-303
Record Dates: First submitted 2021-11-16; First posted 2021-11-26 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: AGA

STUDY DESIGN:
Intervention Model Description: Drug:0.25% (2.275mg/mL) Finasteride Spray Placebo for CU-40102 Spray
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CU-40102 Spray (Experimental): 0.25% (2.275mg/mL) Finasteride
  Interventions: Drug: CU-40102 Spray
- Placebo for CU-40102 Spray (Placebo Comparator): Placebo Spray
  Interventions: Drug: CU-40102 Spray

INTERVENTIONS:
Drug: CU-40102 Spray — topical application, 1~4 sprays each time, once daily

SUMMARY:
A Multicenter, Randomized, Double-Blind, and Placebo-Controlled Phase 3 Clinical Study ,the mean change from baseline in vertex target area hair count (TAHC) after treatment for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Having voluntarily signed the ICF approved by the Ethics Committee and consented to participate in this study before starting any study procedure;
2. Being able to understand and comply with the requirements of the protocol and agreeing to participate in all study visits;
3. Males aged 18 to 41 years (inclusive);
4. Being diagnosed with Type III vertex, Type IV or Type V androgenetic alopecia (AGA) according to the Hamilton-Norwood classification (see Appendix 1 for details);
5. Appropriate medical contraceptive methods being used to prevent the sexual partner from becoming pregnant from the time of signing ICF to 28 days after the last dose; -

Exclusion Criteria:

1. A history of scalp skin abnormalities or scalp skin diseases at the time of screening
2. Patients with secondary alopecia such as those associated with malnutrition, drugs, endocrine , iron deficiency anemia, or systemic lupus erythematosus;
3. Patients with alopecia areata, alopecia cicatrisata, or trichotillomania;
4. Having undergone hair transplantation or extension before screening, or persistent requirement to wear a wig sheath during study treatments;
5. Known allergy to the active ingredient of the investigational drug or any component of the excipients, or to any component of the tattoo liquid;
6. A history of depression, anxiety, personality disorder or other mental disorders;
7. A history of varicocele or infertility ;
8. A history of malignant tumor;

Ages: 18 Years to 41 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
The Rate of TAHC | 24 weeks.
  the change from baseline in target area hair count (TAHC) in the vertex after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People Hosptial, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhou C, Yang B, Zeng H, Xia R, Dang N, Yang Q, Li J, Zhang C, Zhang G, Wei A, Lai W, Yang S, Diao Q, Ding Y, Wu L, Liu L, Jia D, Zhu H, Zhang J. Efficacy and safety of topical finasteride spray solution in the treatment of Chinese men with androgenetic alopecia: A phase III, multicenter, randomized, double-blind, placebo-controlled study. Chin Med J (Engl). 2025 Mar 17. doi: 10.1097/CM9.0000000000003495. Online ahead of print. PMID 40090937